CLINICAL TRIAL: NCT06552065
Title: Comparative Evaluation of Cross-linked Collagen Membrane With and Without Silk Fibroin Around Immediate Dental Implants -Randomized Controlled Trial.
Brief Title: Evaluation of Cross-linked Collagen Membrane With and Without Silk Fibroin Around Immediate Dental Implants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02-D012-00050
Record Dates: First submitted 2024-07-19; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Immediate Implant
Keywords: Silk fibroin with collagen membrane
MeSH Terms: interventions — Collagen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10 will receive cross -linked collagen with silk fibroin membrane around immediate implant. (Experimental): Local anesthesia is given. Atraumatic extraction is done. Osteotomy is done. Immediate implant is placed along with crosslinked collagen with silk fibroin membrane. Suture is done.
  Interventions: Other: collagen with silk fibroin membrane; Other: cross linked collagen membrane
- 10 will receive cross linked collagen membrane around immediate implant (Active Comparator): Local anesthesia is given. Atraumatic extraction is done. Osteotomy is done. Immediate implant is placed along with crosslinked collagen membrane. Suture is done.
  Interventions: Other: collagen with silk fibroin membrane; Other: cross linked collagen membrane

INTERVENTIONS:
Other: collagen with silk fibroin membrane — A mucoperiosteal flap will be raised and atraumatic extraction will be done. An immediate implant with collagen with silk fibroin membrane (experimental group) will be placed according to the standard protocol.
  An immediate implant with collagen membrane ( comparative group) will be placed according to the standard protocol .
  The surgical wound closure will be coapted with mattress and single interrupted sutures
Other: cross linked collagen membrane — A mucoperiosteal flap will be raised and atraumatic extraction will be done. An immediate implant with collagen with silk fibroin membrane (experimental group) will be placed according to the standard protocol.

SUMMARY:
Comparative evaluation of cross-linked collagen membrane with and without silk fibroin around Immediate Dental Implants -Randomized controlled trial.

DETAILED DESCRIPTION:
Periodontal disease is an inflammatory and infectious disease affecting the tooth supporting structures leading to tooth loss when left untreated.The detrimental effect of periodontitis results in soft tissue and hard tissue loss. Bone defects has often resulted from tumor resection, congenital malformation, trauma, fractures, surgery, periodontitis or around implants in dentistry, as well as from diseases, such as osteoporosis or arthritis.These deficiencies have been overcome through various treatment modalities.It is a well-established fact that the cells from the periodontal ligament have the potential for regeneration of the tooth attachment apparatus. In addition, bone grafts and membranes have been used to regenerate the lost bone.

Among the membranes, autogenous connective tissue graft remains as gold standard. Collagen is biocompatible natural polymer that has a good function to promote new tissue formation. In the proposed study, immediate implants with compromised bone support, cross-linked bovine collagen membrane will be used. It is a naturally occurring protein, having excellent biocompatibility, and hemostatic and chemotactic characteristics for gingival fibroblasts and periodontal ligaments. Further, it is resistant to tension, controllable biodegradability, is non cytotoxic, low antigenicity, and excellent anti-inflammatory characteristics. It is naturally reabsorbed by microorganisms, easy to manipulate and has a molecular structure with little variance concerning the animal from which the collagen is extracted, leading to improved immunogenicity.

Bovine collagen is selected to enhance the biological function of silk fibroin, as composite membrane for enhancement of gingival thickness. Thus, considering all these characteristics, silk fibroin is incorporated into collagen membrane for evaluation .As there is no literature assessing this composite membrane, the aim of this study Compare evaluation of Cross-linked collagen membrane with and without Silk fibroin around Immediate Dental Implants Randomized controlled trial will be undertaken.

ELIGIBILITY:
Inclusion Criteria

* Systemically healthy patients in the age group of 18 to 55years.
* Patients undergoing immediate implant placement with gingival thickness ≤ 1mm
* Stage II /Stage III and Grade B Periodontitis patients.
* Radiographic assessment using Radiovisiography (RVG) with grid.

Exclusion Criteria:

* Patients having allergies with collagen and silk products.
* Medical conditions contraindicating surgical interventions.
* Known smokers and alcoholic.
* Acute infections at the site of extraction. Ex Abscess.
* Patients who have undergone radiotherapy or chemotherapy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
To assess wound healing, gingival thickness and keratinized tissue width | pre implant placement , 6 weeks , 12 weeks
  Gingival tissue thickness assessment will be done at the site of implant placement 1.5 mm below the gingival margin of adjacent tooth. Local anaesthesia will be administered before the procedure and an Endodontic K-file with silicone disc stop will be used to measure. The depth will be measured with UNC-15 probe.
  Apico-coronal width of keratinized tissue is measured as the distance from the mucogingival junction to the gingival margin, with the mucogingival junction determined using Schiller's Potassium Iodide Solution.

SECONDARY OUTCOMES:
Radiovisiography with grid | pre implant placement , 6 weeks , 12 weeks
  assess increase in bone volume

CONTACTS AND LOCATIONS:
Locations (1):
- Krishnadevaraya college of dental sciences, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared with other researchers.

REFERENCES:
- [Background] Pripatnanont P, Chankum C, Meesane J, Thonglam J. Physical and biological performances of a semi-resorbable barrier membrane based on silk fibroin-glycerol-fish collagen material for guided bone regeneration. J Biomater Appl. 2021 Nov;36(5):930-942. doi: 10.1177/08853282211025781. Epub 2021 Jun 21. PMID 34152233